CLINICAL TRIAL: NCT03171363
Title: Gaze-Contingent Music Reward Treatment for Anxiety Disorders in Children: A Case Series
Brief Title: Gaze Contingent Feedback for Anxiety Disorders in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor of Psychology and Neuroscience School of Psychological Sciences Sagol School of Neuroscience Tel Aviv University, Tel Aviv University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAUANX
Record Dates: First submitted 2017-05-28; First posted 2017-05-31 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Anxiety Disorders
Keywords: Attention bias modification treatment; Anxiety disorders; Attention training
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gaze-contingent feedback (Experimental): Participants will receive gaze-contingent feedback according to their viewing patterns
  Interventions: Behavioral: Gaze-contingent feedback

INTERVENTIONS:
Behavioral: Gaze-contingent feedback — Participants will receive gaze-contingent feedback according to their viewing patterns

SUMMARY:
The purpose of this study is to determine whether giving gaze-contingent feedback is an effective attention modification procedure, helping in the treatment of anxiety disorders in children.

DETAILED DESCRIPTION:
Attention biases in threat processing have been assigned a prominent role in the etiology and maintenance of anxiety disorders. The purpose of this study is to determine whether giving gaze-contingent feedback is an effective treatment for anxiety disorders in clinically anxious 6-10 year-olds children. Participants will be assessed using clinical interviews and parent- and self-rated questionnaires before and after eight training sessions. Outcome measures will be anxiety symptoms and depression as measured by gold standard questionnaires as well as structured clinical interviews with children and their parents. Attentional threat bias and Attentional control will also be measured to explore potential mediators of ABMT's effect on anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of GAD, SOP, or SAD.
* Co-morbid attention deficit hyperactivity disorder (ADHD) or depressive disorders must be treated with medication and stable.
* Tics or impulse control problems must be treated with medication, stable and cause minimal or no impairment.

Exclusion Criteria: To be excluded youth must:

* meet diagnostic criteria for Organic Mental Disorders, Psychotic Disorders, Pervasive Developmental Disorders, or Mental Retardation.
* show high likelihood of hurting themselves or others.
* have not been living with a primary caregiver who is legally able to give consent for the child's participation.
* be a victim of previously undisclosed abuse requiring investigation or ongoing supervision.
* be involved currently in another psycho-social treatment.
* have a serious vision problem that is not corrected with prescription lenses.
* have a physical disability that interferes with their ability to click a mouse button rapidly and repeatedly.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in anxiety symptoms - the Pediatric Anxiety Rating (PARS) | Post treatment (1 week after treatment completion)
  The PARS assesses global anxiety severity across different anxiety disorders in children

SECONDARY OUTCOMES:
Change from baseline in anxiety related emotional disorders symptoms - Child/Parent (the SCARED 41-item) | Post treatment (1 week after treatment completion)
  The SCARED is a 41-item self and parent-report instrument designed to assess anxiety in children.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No